CLINICAL TRIAL: NCT02043340
Title: Effect of A Single Session Of Antimicrobial Photodynamic Therapy Using Indocyanine Green In The Treatment Of Chronic Periodontitis
Brief Title: Single Session Of Antimicrobial Photodynamic Therapy Using Indocyanine Green
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator, SVS Institute of Dental Sciences
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SVS031102; SVS031102 (Other: Institutional ethics committee, SVSIDS)
Record Dates: First submitted 2014-01-18; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Periodontitis
Keywords: Periodontitis; Bacterial viability; Lactate dehydrogenase levels; Indocyanine green; Scaling and root planing; Antimicrobial photodynamic therapy.
MeSH Terms: conditions — Periodontitis | interventions — Indocyanine Green; Photosensitizing Agents; Lasers; Lasers, Semiconductor; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Indocyanine green (ICG) (Experimental): The study included 30 patients diagnosed with chronic periodontitis. Three sites from three different quadrants were selected and assigned to three groups namely, SRP group - scaling and root planing, LASER group - scaling and root planing with application of 810 nm diode laser and ICG group - scaling and root planing with application of 810 nm diode laser and ICG at a concentration of 5 mg/mL. Primary parameters included estimation of decrease in percentage of viable bacteria at baseline, immediate post treatment and end of 1 week and Lactate dehydrogenase (LDH) levels at baseline and end of 1 week. Secondary parameters included site-specific measures of plaque, gingivitis, pocket depth (PD) and clinical attachment loss (CAL) at specific time intervals.
  Interventions: Drug: indocyanine green; Device: LASER; Procedure: Scaling and Root Planing

INTERVENTIONS:
Drug: indocyanine green — ICG group - scaling and root planing with application of 810 nm diode laser and ICG at a concentration of 5 mg/mL. Primary parameters included estimation of decrease in percentage of viable bacteria at baseline, immediate post treatment and end of 1 week and Lactate dehydrogenase (LDH) levels at baseline and end of 1 week. Secondary parameters included site-specific measures of plaque, gingivitis, pocket depth (PD) and clinical attachment loss (CAL) at specific time intervals.
  Other Names: Cardiogreen; Photosensitizer
Device: LASER — LASER group - scaling and root planing with application of 810 nm diode laser Primary parameters included estimation of decrease in percentage of viable bacteria at baseline, immediate post treatment and end of 1 week and Lactate dehydrogenase (LDH) levels at baseline and end of 1 week. Secondary parameters included site-specific measures of plaque, gingivitis, pocket depth (PD) and clinical attachment loss (CAL) at specific time intervals.
  Other Names: Diode LASER
Procedure: Scaling and Root Planing — SRP group - scaling and root planning. Primary parameters included estimation of decrease in percentage of viable bacteria at baseline, immediate post treatment and end of 1 week and Lactate dehydrogenase (LDH) levels at baseline and end of 1 week. Secondary parameters included site-specific measures of plaque, gingivitis, pocket depth (PD) and clinical attachment loss (CAL) at specific time intervals.
  Other Names: Non-surgical Periodontal Therapy

SUMMARY:
In recent years, there has been a growing interest in the use of dental lasers for treatment of periodontal diseases. Commercially available photodynamic therapy for periodontal diseases utilizes methylene blue as a photosensitizer. In this study, the effects of a novel photosensitizer dye, indocyanine green (ICG), as an adjunct to nonsurgical treatment of chronic periodontitis will be evaluated.

DETAILED DESCRIPTION:
Background and objective: Periodontal disease is caused by periodontal pathogens that colonize the dental plaque and the subsequent host-microbial interactions. The recent years have witnessed a rapid increase in the usage of Light Amplification by Stimulated Emission of Radiation (Laser) in dentistry for the treatment of periodontal diseases. The additive therapeutic effects when a photoactivated dye such as methylene blue is used in conjunction with Laser is well documented. Indocyanine green (ICG), a tri-carbocyanine that belongs to family of cyanine dyes is widely used in the fields of Ophthalmology and Cardiac imaging. Recent in vitro studies have reported its efficacy in killing potent periodontal pathogens like A. actinomycetemcomitans and P. gingivalis when combined with 810 nm diode laser. The present study aims at evaluating the effects of ICG as an adjunct to non-surgical treatment of chronic periodontitis in biofilm environment of human periodontal pockets in terms of immediate reduction in percentage of viable bacteria and at the same to quantitatively assess host tissue injury. Methods: The study included 30 patients diagnosed with chronic periodontitis. Three sites from three different quadrants were selected and assigned to three groups namely, SRP group - scaling and root planing, LASER group - scaling and root planing with application of 810 nm diode laser and ICG group - scaling and root planing with application of 810 nm diode laser and ICG at a concentration of 5 mg/mL. Primary parameters included estimation of decrease in percentage of viable bacteria at baseline, immediate post treatment and end of 1 week and Lactate dehydrogenase (LDH) levels at baseline and end of 1 week. Secondary parameters included site-specific measures of plaque, gingivitis, pocket depth (PD) and clinical attachment loss (CAL) at specific time intervals.

ELIGIBILITY:
Inclusion Criteria:

Patients who were diagnosed with chronic periodontitis having a clinical evidence of periodontal pocket of ≥5mm, in at least 4 sites in each of the 3 quadrants.

* Systemically healthy male & female patients within the age group of 35-55 years.
* No history of medications affecting the periodontium (antibiotics, immunosuppressive drugs, anti-inflammatory, anti-oxidants, antibiotic tooth paste, mouthwashes) or periodontal therapy in the past 24 weeks period leading to the study.

Materials & Methods 26

- Minimum of 5 teeth in each quadrant.

Exclusion Criteria:

Medically compromised patients.

* Patients who had received any antibiotic, periodontal or laser therapy during the past 24 weeks of base line examination.
* Patients using antibacterial mouth rinses or medicated tooth paste during the past 24 weeks.
* Patients with history of tobacco chewing, smoking and alcohol consumption.
* Pregnant women & lactating mothers.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Bacterial Vitality | Baseline to 1 week
  Percentage of viable bacteria were estimated from the subgingival plaque samples at baseline, immediately after treatment and at the end of 1 week using a commercially available bacterial viability kit (LIVE/DEAD® BacLight™ Bacterial Viability Kit, Invitrogen, Leiden, The Netherlands).

SECONDARY OUTCOMES:
LDH | Baseline to 1 week
  LDH activity is used as an indicator of relative cell viability and plasma membrane integrity.,28 Quantitative total LDH was assayed by using a commercially available kit (LDH-Cytotoxicity Assay Kit II (Colorimetric) ®, Abcam, Cambridge, MA, USA). Initially, 10 μL of mammalian cell lysis solution (Cell Lysis Solution, Abcam, Cambridge, MA, USA) was added to every 100 μL of the GCF collected which was subsequently incubated at 30ºC for 5 minutes. The manufacturer's instructions were subsequently followed and the absorbance at 450nm background after subtracting the zero well/NADH background from all readings was recorded by using a colorimetric microplate reader (iMark™ Microplate Absorbance Reader, Bio-Rad, Hyderabad, India). The results are expressed as total LDH activity (mUnits/site) per sample where one unit LDH is the amount of enzyme that catalyzes the conversion of lactate to pyruvate to generate 1.0 μmol to NADH per minute at 37°C.

OTHER OUTCOMES:
Measures of Periodontal Health | Baseline to Six months
  Immediately after the laser application to the LASER group and 0.5 ml of 5mg/ml Indocyanine green dye along with laser to the ICG group by the second operator subgingival plaque samples were collected from the 3 sites by the first operator. The patients were recalled at the end of 1 week for collection of GCF and subgingival plaque samples for the assay of LDH levels and bacterial viability respectively. PI and MGI scores were recorded at the end of 1, 4, 12 and 24 weeks, while PD and CAL were recorded at the end of 12 and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sripriya Nagarajan, MDS, Study Chair — SVS Institute of Dental Sciences